CLINICAL TRIAL: NCT02286817
Title: Phase I Single Dose, Open-label, Pharmacokinetic Study Followed by Single-blind, Placebo-controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Plasma Concentration Profiles, and Targeted Efficacy of NFC-1 in Adolescents (12-17 Years of Age) With Attention-Deficit Hyperactivity Disorder and Genetic Disruption Impacting Metabotropic Glutamate Receptor Genes (NFC1-GREAT)
Brief Title: Phase I Single Dose, Open-Label Pharmacokinetic Study and Single-Blind, Placebo-Controlled Dose Escalation Study of NFC-1 in Adolescents With Attention-Deficit Hyperactivity Disorder
Acronym: NFC1-GREAT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Collaborators: Thomas Jefferson University (Other); Children's Hospital of Philadelphia (Other); Pearson/Clinical Assessment (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFC1-2014
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Attention-deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm of 30 subjects (Experimental): Subjects will be administered single dose of NFC-1 to assess safety, tolerability, and pharmacokinetics, then proceed to continuous, daily administration of NFC-1 for 4 weeks to assess safety, tolerability, and impact on ADHD severity.
  Interventions: Drug: NFC-1

INTERVENTIONS:
Drug: NFC-1 — Single-dose, open label administration to assess safety, tolerability, and pharmacokinetics in adolescents with ADHD and continuous daily administration for four weeks with weekly escalation to evaluate safety, tolerability, and impact on ADHD severity.

SUMMARY:
This trial is a Phase 1 study in adolescents with ADHD and genetic disruptions impacting genes in the metabotropic glutamate receptor (mGluR) network. The objectives of the study are to evaluate the safety, tolerability, and pharmacokinetics following single-dose, oral administration of NFC-1 and to evaluate safety and tolerability and to obtain evidence for the effect of NFC-1 on ADHD severity and global functioning during and following four weeks of continuous treatment. Exploratory analyses will be performed to assess effect size of specific mGluR-network genes on ADHD based on responsiveness of patients to NFC-1. This study will be conducted at a single clinical site, the Jefferson University Hospital PKU (Philadelphia, PA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient's weight is within 5th to 95th percentile for age
2. Patient has ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) and the Vanderbilt ADHD Rating Scale score (Parent or Teacher) > 16 at baseline with or without conventional ADHD therapy
3. Patient has been genotyped (CAP/CLIA certified) to determine whether there are disruptive mutations in genes within the mGluR-network
4. Patient has been a non-smoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months
5. Patient is judged to be in good health, other than having ADHD, based on medical history, physical examination, vital signs measurements, and laboratory safety tests performed at the screening visit and/or prior to administration of study drug
6. Female patients of reproductive potential will have a negative urine β-hCG test at screening and prior to drug administration. If sexually active, female participant agrees to use (and/or have their partner use) two acceptable methods of birth control beginning at least 2 weeks prior to administration of study drug and throughout the study. Acceptable methods of birth control are abstinence, or 2 of the following: intrauterine device (IUD), diaphragm, spermicides, cervical cap, contraceptive sponge, and condoms
7. Patient has no clinically significant abnormality on electrocardiogram (ECG) performed at the screening visit and/or prior to administration of study drug
8. Parent/legal guardian and patient understand the study procedures and agrees to the patient's participation in the study as indicated by parental/legal guardian signature on the patient consent form and patient signature on assent form

Exclusion Criteria:

1. Patient or parent/legal guardian is, in the opinion of the investigator, mentally or legally incapacitated, has significant emotional problems at the time of screening visit or during the conduct of the study. Subjects with prior diagnosis of co-morbid major psychiatric disorders (i.e. aside from ADHD), including major depression, bipolar disease, Tourette syndrome, schizophrenia, autism spectrum disorder or pervasive development disorder, severe anxiety disorders
2. Patient has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the patient by their participation in the study
3. Patient has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Patients with a history of uncomplicated kidney stones may be enrolled in the study at the discretion of the investigator
4. Patient has a history of stroke, chronic seizures, or major neurological disorder
5. Patient is pregnant or a nursing mother
6. Patient has a history of extreme psychological aversion to blood draws that in the opinion of the investigator or parents would result in compromising the study conduct. Patient has a history of extreme physiologic difficulty in venous access that in the opinion of the investigator and parents would result in compromising the study conduct
7. Patient has a history of inability to swallow whole unadulterated pills, which in the opinion of the investigator or parents would result in compromising the study conduct
8. Patient has a systolic or diastolic blood pressure ≥ the 95th percentile for his/her age
9. Patient consumes any alcoholic beverages
10. Patient consumes excessive amounts of caffeine, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day
11. Patient has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription of non-prescription drugs or food
12. Patient is currently a regular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse within approximately 3 years
13. Patient has had surgery, lost more than 5cc/kg of blood, or participated in another investigational drug trial within 4 weeks prior to the screening visit.
14. Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary, or renal disease

    1. AST/SGOT > 2.0 times the upper limit of normal
    2. ALT/SGPT > 2.0 times the upper limit of normal
    3. Total bilirubin > 2.0 times the upper limit of normal
    4. Hemoglobin < 9 gm/dL
    5. White blood cell count < 1,000/ mm3
    6. Platelet count < 100,000/mm3
15. Any investigational drug use within 30 days prior to enrollment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Assessing the safety and tolerability of NFC-1 at each dose level based on assessment of adverse events and other safety measurements including vital signs, electrocardiogram, laboratory safety tests. | 24 hours
Profile pharmacokinetics of NFC-1 in adolescents when administered orally as single dose. | 24 hours
Assessing the safety and tolerability of NFC-1 during 4 weeks of continuous daily administration based on assessment of adverse events and other safety measurements including vital signs, electrocardiogram, laboratory safety tests. | 1-4 weeks

SECONDARY OUTCOMES:
The change in Vanderbilt scores during and following 4-week treatment with NFC-1 | 1-4 weeks
The change in Actigraphy scores during and following 4-week treatment with NFC-1 | 1-4 weeks
The change in Quotient ADHD test scores during and following 4-week treatment with NFC-1 | 1-4 weeks
The change in PERMP-MATH test scores during and following 4-week treatment with NFC-1 | 1-4 weeks
The change in Clinical Global Impressions Severity/Improvement scores during and following 4-week treatment with NFC-1 | 1-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kraft, MD, Principal Investigator — Thomas Jefferson University; Josephine Elia, MD, Principal Investigator — Alfred I. duPont Hospital for Children
Locations (1):
- Thomas Jefferson University, Clinical Research Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glessner JT, Khan ME, Chang X, Liu Y, Otieno FG, Lemma M, Slaby I, Hain H, Mentch F, Li J, Kao C, Sleiman PMA, March ME, Connolly J, Hakonarson H. Rare recurrent copy number variations in metabotropic glutamate receptor interacting genes in children with neurodevelopmental disorders. J Neurodev Disord. 2023 Apr 29;15(1):14. doi: 10.1186/s11689-023-09483-z. PMID 37120522
- [Derived] Slaby I, Hain HS, Abrams D, Mentch FD, Glessner JT, Sleiman PMA, Hakonarson H. An electronic health record (EHR) phenotype algorithm to identify patients with attention deficit hyperactivity disorders (ADHD) and psychiatric comorbidities. J Neurodev Disord. 2022 Jun 11;14(1):37. doi: 10.1186/s11689-022-09447-9. PMID 35690720
- [Derived] Elia J, Ungal G, Kao C, Ambrosini A, De Jesus-Rosario N, Larsen L, Chiavacci R, Wang T, Kurian C, Titchen K, Sykes B, Hwang S, Kumar B, Potts J, Davis J, Malatack J, Slattery E, Moorthy G, Zuppa A, Weller A, Byrne E, Li YR, Kraft WK, Hakonarson H. Fasoracetam in adolescents with ADHD and glutamatergic gene network variants disrupting mGluR neurotransmitter signaling. Nat Commun. 2018 Jan 16;9(1):4. doi: 10.1038/s41467-017-02244-2. PMID 29339723